CLINICAL TRIAL: NCT06203041
Title: Vitamin D Sulfates in Breastmilk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas Thacher, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-005324
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Vitamin D Deficiency; Breast Milk Collection
MeSH Terms: conditions — Vitamin D Deficiency; Breast Milk Expression | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactating women (Experimental): Subjects identified as having delivered an infant and lactating will receive Vitamin D3 for 28 days.
  Interventions: Dietary Supplement: Vitamin D
- Breastfeeding Infants (No Intervention): No intervention will be administered.

INTERVENTIONS:
Dietary Supplement: Vitamin D — Orally administered, daily dose of 5000 IU (125 mcg) Vitamin D3 for 28 days.
  Other Names: cholecalciferol
  Arms: Lactating women

SUMMARY:
Infants The purpose of this study is to measure breastmilk's vitamin D sulfate nutritional value in infant's saliva and digesta (gut).

Breastfeeding Mothers The purpose of this study is to measure Vitamin D sulfates in freshly expressed breastmilk samples before and after 28 days of Vitamin D supplementation in lactating mothers.

DETAILED DESCRIPTION:
Infants

Sign the consent form to confirm participation:

You will be asked to bring a soiled diaper from the morning of the study visit. You will meet with a study team member who will collect up to 6 swabs total:

Up to 3 cheek/mouth swabs to collect saliva Up to 3 stool/anus/diaper swabs

Lactating Mothers

Sign the consent form to confirm participation:

Visit 1 (Baseline) You will meet with a study team member complete some demographic information and gestational age of the baby and birthdate, next you will have a blood draw and express breast milk in a private location, the study team will collect up to 50 ml of freshly expressed breast milk for the research study, you will be asked to bring your personal breast pump and collection container to each research visit, or manually express milk, see options below. The study team member will schedule visit 2. The study will provide the vitamin D supplement that you will take daily for 28 days.

Visit 2 (post intervention) Approximately 28 days later you will meet with a study team member, have a blood draw and express breast milk in a private location, the study team will collect up to 50 ml of freshly expressed breast milk for the research study, you will be asked to bring your personal breast pump and collection container to each research visit, or manually express milk, see options below. The study team member will ask for the container the Vitamin D supplement was in.

You have 2 options:

Option 1:

Bring along your personal breast pump and collection container to each study visit.

The study team member will collect up to 50 ml of freshly expressed breast milk for the study.

Option 2:

You do not bring along your personal breast pump and containers to each study visit, instead you will be asked to:

Manually express your breast milk into a specimen collection cup at each study visit.

ELIGIBILITY:
Lactating Mothers

Inclusion Criteria:

* Lactating mothers
* ≥2 weeks after delivery
* No intentions of weaning during the study

Exclusion Criteria:

* History of sarcoidosis
* History of renal disease
* Premature birth- <37 weeks
* Taking daily supplement with ≥600 IU vitamin D in the past 30 days

Breastfeeding Infants

Inclusion Criteria:

* Female and male infants
* Exclusively breastfed

Exclusion Criteria:

* No known gastrointestinal diseases that require medical treatment
* Currently prescribed antibiotics or have taken antibiotics <2 weeks from collection

Ages: 1 Month to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Vitamin D sulfate levels in breastmilk | Baseline, Day 28
  Samples will be assessed using a Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) assay on the Agilent 6490 tandem mass spectrometer instrument.

SECONDARY OUTCOMES:
Vitamin D sulfate levels in infant saliva | Baseline
  Samples will first be assessed for activity using a general sulfatase activity assay, followed by a Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) assay on the Agilent 6490 tandem mass spectrometer instrument.
Vitamin D sulfate levels in infant digesta | Baseline
  Samples will first be assessed for activity using a general sulfatase activity assay, followed by a Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) assay on the Agilent 6490 tandem mass spectrometer instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Thatcher, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials